CLINICAL TRIAL: NCT05094557
Title: Clinical Efficacy of a Virtual Reality Tool for the Treatment of Obesity (SOCRATES)
Brief Title: Clinical Efficacy of a Virtual Reality Tool for the Treatment of Obesity
Acronym: SOCRATES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOCRATES_RCT/2021; 951930 (Other Grant/Funding Number: Horizon 2020)
Record Dates: First submitted 2021-09-27; First posted 2021-10-26 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Obesity, Morbid
Keywords: Virtual Reality; obesity; Motivational Interviewing; embodiment; psychological treatment
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): Participants from the Experimental Group 1 will engage in a self-conversation through embodied perspective taking (body swapping), according to which they will be embodied alternately in their own virtual representation and in their counsellor's virtual body. They will also continue receiving Treatment As usual plus a Psychoeducational video with useful information about how to engage with a healthier lifestyle.
  Interventions: Behavioral: Experimental Group 1: Body swapping VR intervention + psychoeducational video + Treatment As usual
- Experimental Group 2 (Experimental): Participants from the Experimental Group 2 will be embodied in their own body and will participate in a "pre-established discourse" provided by their virtual counsellor. Participants will also continue receiving Treatment As usual plus a Psychoeducational video with useful information about how to engage with a healthier lifestyle.
  Interventions: Behavioral: Experimental Group 2: VR intervention without body swapping + psychoeducational video + Treatment As usual
- Control Group (Active Comparator): Participants from the Control Group will receive their Treatment As Usual plus a Psychoeducational video. Treatment as usual will consist of regular medical, nutritional and/or psychiatric follow-ups with the obesity specialists of the Vall d´ Hebron University Hospital and standard routine tests. These visits aim to provide practical recommendations about how to achieve a gradual weight loss and engage more with physical exercise.
  Interventions: Behavioral: Control Group: Psychoeducational video + Treatment As usual

INTERVENTIONS:
Behavioral: Experimental Group 1: Body swapping VR intervention + psychoeducational video + Treatment As usual — The patient will be embodied in his/her own avatar and will maintain a conversation with a counsellor's avatar of his/her choice. Once the experiment starts, the patient, embodied in his/her own body, will start describing his/her problem in terms of subjective experiences of being obese in daily life. Then, he/she will be body swapped to the counsellor's body and try to respond to the problem just manifested by the patient. The crucial aspect here is that the patient, from the counsellor's viewpoint, will see a representation of his/her real body when looking at the patient's avatar speaking and moving. Therefore, the patient will have the opportunity to see himself/herself in first person (1PP) and second person (2PP) perspectives.
  Other Names: EG1
  Arms: Experimental Group 1
Behavioral: Experimental Group 2: VR intervention without body swapping + psychoeducational video + Treatment As usual — Participants from the Experimental Group 2 will be embodied in their own body and will participate in "pre-established discourse" provided by the chosen counsellor, who will ask about the perceived barriers for engagement with a healthier lifestyle and will give practical recommendations about how to achieve a healthier and happier life, in terms of healthy eating and physical activity. No body swapping will take place for this group. Participants will also continue receiving Treatment As usual plus a Psychoeducational video with useful information about how to engage with a healthier lifestyle.
  Other Names: EG2
  Arms: Experimental Group 2
Behavioral: Control Group: Psychoeducational video + Treatment As usual — Participants from the Control Group will receive their Treatment As Usual plus a Psychoeducational video. Treatment as usual will consist of regular medical, nutritional and/or psychiatric follow-ups with the obesity specialists of the Vall d´ Hebron University Hospital and standard routine tests. These visits aim to provide practical recommendations about how to achieve a gradual weight loss and engage more with physical exercise.
  Other Names: CG
  Arms: Control Group

SUMMARY:
The objective of the study, which is framed within European Union's H2020 project titled SOCRATES, is to assess the clinical efficacy of a Virtual Reality (VR) embodiment tool for treating obesity and to compare it to usual care, through a Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 and ≤ 55 kg/m2.
* Receiving ambulatory treatment at the Vall d´Hebron University Hospital.
* No concurrent involvement in other treatment related to the obesity condition.
* Minimal digital skills and able to use a proper digital device (Smartphone, tablet, computer).
* Oral and written understanding of the Spanish language to complete the questionnaires and use the system.
* Acceptance to sign the informed consent to participate.

Exclusion Criteria:

* Body Mass Index > 45.
* Presence of an Eating Disorder during the last 2 years.
* Non-stabilised severe mental disorder that could interfere with the successful implementation of the research protocol (i.e. psychosis, depression with suicidal risk, alcohol or drug abuse, psychotic or manic symptoms).
* Auditory or visual complications that might affect the participant during exposure to the VR platform.
* Intellectual disability or any major illness seriously affecting cognitive performance (i.e. neurological disorders).
* Personal history of epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Readiness to change I | Baseline (week 0); Post-Experiment1 (week 3)- Baseline; Post-Experiment2 (week 4)- Baseline; Post-Experiment3 (week 5) - Baseline; Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Readiness Rulers are Visual Analogue Scales ranging from 1 to 10 that assess "Importance", "Confidence" and "Readiness" to change. For the present study, these 3 variables will be measured in terms of a) achieving a healthy weight and b) exercising more, while the "Readiness" scale will be used as critical response primary variable.
Readiness to change II | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  As a complementary readiness to change measure, the Spanish version of the Stages of Change in Overweight and Obese People (S-Weight) and the Processes of Change in Overweight and Obese People (P-Weight) will be used. Regarding P-Weight, lower scores on this scale reflect no use of a given process of change and higher scores reflect the full use of that process. To make scores from the different subscales comparable, these scores are transformed on a scale ranging from 0 to 100.

SECONDARY OUTCOMES:
Eating habits I | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Three Factor Eating Questionnaire-R18 (TFEQ-R18). The questionnaire assesses three different aspects of eating behaviour: (a) cognitive restraint (CR); (b) uncontrolled eating (UE) and (c) emotional eating (EE). The questionnaire consists of 18 items using a 4-point response scale which ranges from 1 (definitely true) to 4 (definitely false) and items scores are summated into the 3 different subscales: CR, UE and EE. Lower scores show more disordered eating while higher scores show healthier eating behaviour.
Eating habits II | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Lifestyle habits questionnaire. The questionnaire consists of 22 items, each one of which is rated using a 5-poing Likert scale ranging from 1 (Never) to 5 (always), with higher scores indicated better lifestyle habits.
Psychological well-being I | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Hamilton Anxiety and Depression Scale (HADS). The questionnaire consists of 14 items, 7 for anxiety and 7 for depression, and is used to detect the presence and severity of anxiety and depression among people with physical illnesses. The HADS is scored on a 4-point Likert scale ranging from 0 to 3, with the total score ranging from 0 to 42. Higher scores indicate a greater level of distress.
Psychological well-being II | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Body Shape Questionnaire (BSQ). The BSQ is a 10-item self-report instrument, derived from the original 34-item version developed by Cooper, Taylor, Cooper, & Fairbum (1987), which assesses concerns about body shape expressed by clinical and non-clinical samples. It is based on a 6-point Likert scale questions (Never, Rarely, Sometimes, Often, Very Often, and Always) with higher scores indicating higher body dissatisfaction.
Psychological well-being III | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Body Image QoL Inventory (BIQLI-SP). The BIQLI is a 19-item instrument designed to quantify the impact of one's body image experiences on several relevant facets of his/her psychosocial functioning and wellbeing in everyday life. The instrument uses a 7-point bipolar scale ranging from -3 (very negative effect) to 0 (no impact) to +3 (very positive impact), with higher scores indicating better psychological well-being in everyday life.
Psychological well-being IV | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Weight Bias Internalization Scale (WBIS-M). The WBIS-M is a self-report 11-item unidimensional scale that is considered one of the most frequently used instruments for assessing internalized weight stigma across different body weight categories, in both clinical and research settings. Each answer is rated using a 7-point Liker scale, ranging from 1 (Strongly disagree) to 7 (Strongly agree) with higher scores indicating higher internalized weight bias. Items 1 and 9 are reverse scored.
Body Mass Index | Baseline (week 0); Post-Intervention (week 6)- Baseline; 1-week follow-up (week 7)- Baseline; 4-week follow-up (week 10)- Baseline
  Body Mass Index (kg/m2)
Cognitive Reserve Questionnaire | Baseline (week 0)
  The CRQ is a self-report questionnaire developed and validated in Spanish population, which evaluates the degree of Cognitive Reserve (CR) in healthy controls and in patients with early signs of Alzheimer disease. The CRQ is composed of 8 items that assess aspects generally related to cognitive reserve ranges from 0 to 25 and is divided into quartiles. In this way, a score equal to or less than 6 points (≤ Q1) would show a low CR, between 7 and 9 points (Q1-Q2) would correspond to a low-medium CR, while scores between 10 and 14 (Q2-Q3) would show medium-high CR. Finally, scores ≥ 15 points would be classified as high CR (Q4).

OTHER OUTCOMES:
Adherence and satisfaction with the VR platform I | Post-Experiment1 (week 3); Post-Experiment2 (week 4)- Post-Experiment1; Post-Experiment3 (week 5)- Post-Experiment1; Post-Intervention (week 6)- Post-Experiment1
  Suitability Evaluation Questionnaire (SEQ). The SEQ is a 14-item questionnaire designed to measure satisfaction, acceptance and security of use in VR systems and it was specifically designed for rehabilitation systems using VR. Thirteen questions of the SEQ are based on a 6-point Likert scale plus a last open-ended question offering participants the possibility to add comments, if necessary. The global score of SEQ ranges from 13 (poor suitability) to 65 (excellent suitability).
Adherence and satisfaction with the VR platform II | Post-Experiment1 (week 3); Post-Experiment2 (week 4)- Post-Experiment1; Post-Experiment3 (week 5)- Post-Experiment1; Post-Intervention (week 6)- Post-Experiment1
  Body Ownership questionnaire does a subjective rating of the illusion of body ownership during the virtual experience through 4 questions that use a 7-point Likert scale, where -3 means "not at all" and +3 "very much" (1. body ownership when looking down; 2. body ownership when looking at the mirror; 3. body ownership when moving; 4. self recognition).
Adherence and satisfaction with the VR platform III | Post-Experiment1 (week 3); Post-Experiment2 (week 4); Post-Experiment3 (week 5); Post-Intervention (week 6)
  User experiment and feedback (qualitative / interview)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Lusilla-Palacios, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Psychiatry Department; Vall d'Hebron Institute of Research, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author once the study is published. The data are not publicly available due to the sensitivity of participants´data.

REFERENCES:
- [Derived] Anastasiadou D, Herrero P, Garcia-Royo P, Vazquez-De Sebastian J, Slater M, Spanlang B, Alvarez de la Campa E, Ciudin A, Comas M, Ramos-Quiroga JA, Lusilla-Palacios P. Assessing the Clinical Efficacy of a Virtual Reality Tool for the Treatment of Obesity: Randomized Controlled Trial. J Med Internet Res. 2024 Apr 5;26:e51558. doi: 10.2196/51558. PMID 38578667
- [Derived] Anastasiadou D, Slater M, Spanlang B, Cano Porras D, Comas M, Ciudin A, Puig GP, Vazquez-De Sebastian J, Ramos-Quiroga JA, Lusilla-Palacios P. Clinical efficacy of a virtual reality tool for the treatment of obesity: study protocol of a randomised controlled trial. BMJ Open. 2022 Jun 22;12(6):e060822. doi: 10.1136/bmjopen-2022-060822. PMID 35732390